CLINICAL TRIAL: NCT04409457
Title: The Influences of Eating and Fasting on Inhibitory Control in Bulimia Nervosa: A Computational Neuroimaging Study
Brief Title: Self-Control in Bulimia Nervosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Laura Berner, Associate Professor of Psychiatry, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: GCO 19-1047; K23MH118418 (NIH)
Record Dates: First submitted 2020-05-18; First posted 2020-06-01 (Actual); Results first posted 2026-01-14 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-11

CONDITIONS: Bulimia Nervosa
Keywords: bulimia nervosa; binge eating; purging; fasting; eating disorder; control
MeSH Terms: conditions — Bulimia Nervosa; Bulimia; Fasting; Feeding and Eating Disorders | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: Two participant groups (one with and one without bulimia nervosa) will be scanned using MRI after they have fasted and after they have consumed a standardized meal. The order of these two scans will be counterbalanced across groups.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants with Bulimia Nervosa (Other): Participants are randomly assigned (in even numbers across the two groups) to scan order:
  A. These participants are first scanned after 16 hours of fasting on one day, and are next scanned after a standardized meal on a second day.
  B. These participants are first scanned after a standardized meal on one day, and are next scanned after 16 hours of fasting on a second day.
  Interventions: Other: fasting state; Other: fed state; Other: magnetic resonance imaging
- Participants without Bulimia Nervosa (Other): Participants are randomly assigned (in even numbers across the two groups) to scan order:
  A. These participants are first scanned after 16 hours of fasting on one day, and are next scanned after a standardized meal on a second day.
  B. These participants are first scanned after a standardized meal on one day, and are next scanned after 16 hours of fasting on a second day.
  Interventions: Other: fasting state; Other: fed state; Other: magnetic resonance imaging

INTERVENTIONS:
Other: fasting state — 16 hours of fasting
Other: fed state — fed a standardized meal
Other: magnetic resonance imaging — neuroimaging with computational modeling
  Other Names: MRI

SUMMARY:
This study examines the influence of acute fasting and eating on self-control in adult females with and without bulimia nervosa (BN). Specifically, the study team is investigating whether differences in behavior and brain activation in response to computer tasks after fasting and after eating a meal could help to explain the symptoms of bulimia nervosa. Data will be collected using questionnaires and a technology called magnetic resonance imaging (MRI).

DETAILED DESCRIPTION:
Treatment-resistant binge eating and purging may be perpetuated by self-control deficits linked to reduced activation in frontostriatal circuits. To date, however, neurocognitive studies of BN have not assessed the dynamic computational processes underlying inhibition or considered the fact that individuals with BN oscillate between two extremes-under-controlled and over-controlled intake. The proposed study combines neuroimaging with computational modeling to investigate the influences of acute fasting and eating (i.e., metabolic states) on how the brains of women with bulimia nervosa (BN) adaptively prepare for and exert inhibitory control. More specifically, the study has the following main objectives: 1) To determine whether eating and fasting affect adaptive inhibitory control and related frontostriatal activation abnormally in BN; 2) To identify associations of BN severity with state-specific frontostriatal activation and behavior.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 18 to 35 years
* Currently between 85 and 130% of the expected weight for height
* Right-handed
* English-speaking

Additional Inclusion Criteria for Women with Bulimia Nervosa:

- Meet DSM-5 criteria for bulimia nervosa

Exclusion Criteria:

* Medical instability
* Ongoing medical treatment, medical condition, or psychiatric disorder that may interfere with study variables or participation
* Shift work
* Pregnancy, planned pregnancy, or lactation during the study period
* Allergy to any of the ingredients in or unwillingness to consume the standardized meal or unwillingness to drink water during the fasting period
* Any contraindication for fMRI

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The prevalence of bulimia nervosa is substantially greater in women than in men. Moreover, prior research suggest that men and women show different neural response patterns during the engagement of inhibitory control, and that satiety differentially impacts the neural function of men and women.
Enrollment: 100 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2024-11-05 (Actual); Study Completion 2024-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura A Berner, PhD, Principal Investigator — Department of Psychiatry, Icahn School of Medicine at Mount Sinai
Locations (1):
- Center of Excellence in Eating and Weight Disorders at the Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: SAP
Time Frame: Beginning 24 months following peer-reviewed article publication
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 100 individuals were recruited (from New York City and the surrounding community and the Center of Excellence in Eating and Weight Disorders at Mount Sinai) and signed informed consent for the full study.
Pre-assignment Details: Subjects completed several screening processes to determine eligibility.
Groups:
- Participants With Bulimia Nervosa: Participants with Bulimia Nervosa who signed consent
- Healthy Control Participants Without Bulimia Nervosa: Healthy Control Participants without Bulimia Nervosa who signed consent
- Bulimia Nervosa Fast Then Fed: Participants were scanned after 16 hours of fasting (Fasted Scan) on one day, and were scanned after a standardized meal on a separate day (Fed Scan).
- Bulimia Nervosa Fed Then Fast; Healthy Control Fed Then Fast: Participants are scanned after a standardized meal on one day (Fed Scan) and are scanned after 16 hours of fasting (Fasted Scan) on a separate day,
- Healthy Control Fast Then Fed: Participants are scanned after 16 hours of fasting (Fasted Scan) on one day, and are scanned after a standardized meal on a separate day (Fed Scan).
Period: Screening Prior to Randomization
Arm/Group | Participants With Bulimia Nervosa | Healthy Control Participants Without Bulimia Nervosa | Bulimia Nervosa Fast Then Fed | Bulimia Nervosa Fed Then Fast | Healthy Control Fast Then Fed | Healthy Control Fed Then Fast
Started | 51 | 49 | 0 | 0 | 0 | 0
Completed | 33 | 35 | 0 | 0 | 0 | 0
Not Completed | 18 | 14 | 0 | 0 | 0 | 0
Not completed — Screening fail prior to randomization | 16 | 13 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 0 | 0 | 0
Period: Randomization
Arm/Group | Participants With Bulimia Nervosa | Healthy Control Participants Without Bulimia Nervosa | Bulimia Nervosa Fast Then Fed | Bulimia Nervosa Fed Then Fast | Healthy Control Fast Then Fed | Healthy Control Fed Then Fast
Started | 0 | 0 | 16 | 17 | 18 | 17
Completed | 0 | 0 | 16 | 16 | 17 | 15
Not Completed | 0 | 0 | 0 | 1 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Incidental MRI finding at scan 1 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Technical/equipment error at scan 1 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Participants With Bulimia Nervosa; Healthy Control Participants Without Bulimia Nervosa: Participants were scanned after 16 hours of fasting (Fasted Scan) on one day, and were scanned after a standardized meal on a separate day (Fed Scan). The order of these fasted and fed visits was counterbalanced across participants.
- Total: Total of all reporting groups
Arm/Group | Participants With Bulimia Nervosa | Healthy Control Participants Without Bulimia Nervosa | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.00 (4.64) | 24.88 (3.65) | 24.94 (4.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 32 | 64
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 25 | 51
  Not Hispanic or Latino | 6 | 7 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 11 | 12 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 6 | 8
  White | 14 | 10 | 24
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 4 | 3 | 7
Number of objective binge eating episodes [Mean (Standard Deviation); unit: episodes in past 28 days] — Eating Disorder Examination (EDE): Frequency of objective binge eating episodes - number of times the behavior occurred (past 28 days) Population: For healthy controls, EDE was administered to confirm healthy control status. Data not relevant in healthy controls, who by definition could not have any binge eating.
  episodes in past 28 days
    Participants with Bulimia Nervosa: number analyzed (Participants) | 32 | 0 | 32
    Participants with Bulimia Nervosa | 12.7 (11.4) |  | 12.7 (11.4)
    Healthy Control: number analyzed (Participants) | 0 | 32 | 32
    Healthy Control |  | 0 (0) | 0 (0)
Number of self-induced vomiting episodes [Mean (Standard Deviation); unit: number of episodes in the past 28 days] — EDE: Frequency of self-induced vomiting episodes - number of times the behavior occurred (past 28 days). Population: For healthy controls, EDE was administered to confirm healthy control status. Data not relevant in healthy controls, who by definition could not have any purging behaviors.
  number of episodes in the past 28 days
    Participants with Bulimia Nervosa: number analyzed (Participants) | 32 | 0 | 32
    Participants with Bulimia Nervosa | 10.2 (13.1) |  | 10.2 (13.1)
    Healthy Control: number analyzed (Participants) | 0 | 32 | 32
    Healthy Control |  | 0 (0) | 0 (0)
Number of fasting episodes [Mean (Standard Deviation); unit: number of episodes in the past 28 days] — EDE: Frequency of fasting episodes - number of times the behavior occurred (past 28 days) Population: For healthy controls, EDE was administered to confirm healthy control status. Data not relevant in healthy controls, who by definition could not have any fasting episodes.
  number of episodes in the past 28 days
    Participants with Bulimia Nervosa: number analyzed (Participants) | 32 | 0 | 32
    Participants with Bulimia Nervosa | 8.69 (7.75) |  | 8.69 (7.75)
    Healthy Control: number analyzed (Participants) | 0 | 32 | 32
    Healthy Control |  | 0 (0) | 0 (0)

OUTCOME MEASURES:

1. Primary Outcome: Brain Activation Associated With P(Stop)
Description: Frontostriatal activation modulated by the predicted need for inhibition (P(stop) (i.e., parametric modulation by p(Stop)), measured as the mean BOLD signal across voxels within the region of interest (ROI). Positive values indicate that neural activation increases as the predicted probability of needing to stop increases (i.e., stronger responses when stopping is predicted to be more likely), whereas negative values indicate that activation decreases as the predicted probability of needing to stop increases (i.e., greater activation when stopping is predicted to be less likely).
Time Frame: after 16 hours of fasting and at 30 minutes after a standardized meal (as least 24 hours apart, but not more than 7 days apart)
Population: Brain imaging data were pre-processed and analyzed for each group and state. Data from 8 participants were excluded: 2 HC due to technical malfunction that caused loss of behavioral data from their 2nd MRI visit, 1 HC for incidental finding on MRI (not identified until after their 2nd scan), 2 (1 BN, 1 HC) for insufficient trials for analysis in a key condition at one or both scans, and 3 BN for excessive movement (>20% of TRs with ≥0.5mm framewise displacement) at one or both scans.
Measure: Mean (Standard Deviation); unit: BOLD Signal
Groups:
- Participants With Bulimia Nervosa (Fasted Scan); Healthy Control Participants (Fasted Scan): Participants are scanned after 16 hours of fasting (Fasted Scan)
- Participants With Bulimia Nervosa (Fed Scan); Healthy Control Participants (Fed Scan): Participants are scanned after a standardized meal (Fed Scan).
Arm/Group | Participants With Bulimia Nervosa (Fasted Scan) | Participants With Bulimia Nervosa (Fed Scan) | Healthy Control Participants (Fasted Scan) | Healthy Control Participants (Fed Scan)
Number analyzed (Participants) | 28 | 28 | 28 | 28
BOLD Signal
  Left DLPFC Brain Activation | 0.02 (0.32) | 0.11 (0.35) | 0.04 (0.41) | 0.05 (0.34)
  Left Caudate Brain Activation | -0.16 (0.36) | -0.06 (0.35) | -0.05 (0.31) | -0.07 (0.39)
  Left Putamen Brain Activation | -0.06 (0.28) | -0.01 (0.27) | 0.02 (0.31) | -0.01 (0.29)
  Left Dorsal ACC Activation | -0.07 (0.27) | 0 (0.29) | -0.08 (0.30) | -0.06 (0.31)
  Left VLPFC Brain Activation | 0.01 (0.28) | 0.03 (0.29) | -0.01 (0.32) | 0.02 (0.28)
  Right DLPFC Brain Activation | 0.07 (0.36) | 0.14 (0.37) | 0.14 (0.36) | 0.12 (0.34)
  Right Caudate Brain Activation | -0.12 (0.42) | 0 (0.38) | -0.02 (0.32) | -0.01 (0.45)
  Right Putamen Brain Activation | -0.05 (0.31) | -0.01 (0.29) | 0.02 (0.35) | -0.01 (0.30)
  Right Dorsal ACC Activation | -0.07 (0.25) | 0 (0.23) | -0.05 (0.26) | -0.04 (0.29)
  Right VLPFC Brain Activation | 0.01 (0.33) | 0.02 (0.24) | 0.03 (0.29) | -0.01 (0.27)

2. Primary Outcome: Brain Activation Associated With Prediction Errors (Unsigned)
Description: Frontostriatal activation modulated by unsigned inhibitory control prediction errors (i.e., parametric modulation by absolute prediction error magnitude), measured as the mean BOLD signal across voxels within the region of interest (ROI). Positive values indicate that neural activation increases with the magnitude of unsigned prediction errors (i.e., stronger responses to more surprising outcomes), whereas negative values indicate that activation decreases as unsigned prediction errors increase (i.e., relative deactivation for more surprising outcomes).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: BOLD Signal
Arm/Group | Participants With Bulimia Nervosa (Fasted Scan) | Participants With Bulimia Nervosa (Fed Scan) | Healthy Control Participants (Fasted Scan) | Healthy Control Participants (Fed Scan)
Number analyzed (Participants) | 28 | 28 | 28 | 28
BOLD Signal
  Left DLPFC Brain Activation | 0.09 (0.29) | 0.13 (0.35) | 0.08 (0.40) | 0.09 (0.29)
  Left Caudate Brain Activation | 0.07 (0.35) | 0.11 (0.30) | 0.06 (0.46) | 0.08 (0.32)
  Left Putamen Brain Activation | -0.03 (0.26) | -0.02 (0.32) | 0.01 (0.35) | -0.06 (0.39)
  Left Dorsal ACC Activation | -0.02 (0.32) | 0.07 (0.29) | 0.09 (0.41) | -0.01 (0.26)
  Left VLPFC Brain Activation | 0.04 (0.31) | 0.11 (0.36) | 0.09 (0.40) | 0.04 (0.26)
  Right DLPFC Brain Activation | 0.33 (0.37) | 0.32 (0.31) | 0.38 (0.38) | 0.39 (0.36)
  Right Caudate Brain Activation | 0.12 (0.38) | 0.12 (0.29) | 0.07 (0.53) | 0.14 (0.32)
  Right Putamen Brain Activation | 0.13 (0.31) | 0.08 (0.28) | 0.14 (0.35) | 0.07 (0.35)
  Right Dorsal ACC Activation | 0.05 (0.28) | 0.10 (0.25) | 0.09 (0.35) | 0.01 (0.24)
  Right VLPFC Brain Activation | 0.29 (0.26) | 0.28 (0.23) | 0.45 (0.30) | 0.34 (0.30)

3. Primary Outcome: Brain Activation Associated With Prediction Errors (Signed)
Description: Frontostriatal activation modulated by signed inhibitory control prediction errors (i.e., parametric modulation by prediction error magnitude), measured as the mean BOLD signal across voxels within the region of interest (ROI). Positive values indicate that neural activation increases as signed prediction errors become more positive (i.e., stronger responses to the surprising need for control), whereas negative values indicate that activation decreases as signed prediction errors become more positive (i.e., stronger responses to the surprising lack of need for control).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: BOLD Signal
Arm/Group | Participants With Bulimia Nervosa (Fasted Scan) | Participants With Bulimia Nervosa (Fed Scan) | Healthy Control Participants (Fasted Scan) | Healthy Control Participants (Fed Scan)
Number analyzed (Participants) | 28 | 28 | 28 | 28
BOLD Signal
  Left DLPFC Brain Activation | 0.05 (0.29) | 0.07 (0.40) | 0.03 (0.40) | 0.02 (0.32)
  Left Caudate Brain Activation | 0.16 (0.35) | 0.16 (0.34) | 0.06 (0.45) | 0.05 (0.41)
  Left Putamen Brain Activation | -0.04 (0.25) | -0.07 (0.33) | -0.07 (0.34) | -0.13 (0.41)
  Left Dorsal ACC Activation | 0.03 (0.36) | 0.09 (0.36) | 0.10 (0.43) | -0.01 (0.31)
  Left VLPFC Brain Activation | 0.02 (0.33) | 0.10 (0.41) | 0.07 (0.39) | 0.03 (0.26)
  Right DLPFC Brain Activation | 0.25 (0.33) | 0.24 (0.36) | 0.28 (0.39) | 0.30 (0.38)
  Right Caudate Brain Activation | 0.15 (0.37) | 0.09 (0.36) | 0.04 (0.48) | 0.10 (0.40)
  Right Putamen Brain Activation | 0.12 (0.29) | 0.06 (0.28) | 0.06 (0.33) | 0.02 (0.40)
  Right Dorsal ACC Activation | 0.09 (0.31) | 0.11 (0.32) | 0.11 (0.36) | 0.02 (0.28)
  Right VLPFC Brain Activation | 0.28 (0.27) | 0.29 (0.27) | 0.44 (0.31) | 0.36 (0.32)

4. Primary Outcome: Brain Activation Associated With Successful Inhibition
Description: Frontostriatal activation associated with successful inhibition , measured as the mean BOLD signal across voxels within the region of interest (ROI) for the contrast of Successful Stop vs. Go trials. Positive values indicate activation associated with successful inhibition.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: BOLD Signal
Arm/Group | Participants With Bulimia Nervosa (Fasted Scan) | Participants With Bulimia Nervosa (Fed Scan) | Healthy Control Participants (Fasted Scan) | Healthy Control Participants (Fed Scan)
Number analyzed (Participants) | 28 | 28 | 28 | 28
BOLD Signal
  Left DLPFC Brain Activation | 0.06 (0.27) | 0.11 (0.40) | 0.08 (0.36) | 0.06 (0.33)
  Left Caudate Brain Activation | 0.18 (0.30) | 0.21 (0.31) | 0.12 (0.48) | 0.10 (0.36)
  Left Putamen Brain Activation | 0.06 (0.23) | 0.09 (0.33) | 0.07 (0.37) | 0.04 (0.39)
  Left Dorsal ACC Activation | -0.04 (0.32) | 0.09 (0.37) | 0.06 (0.43) | -0.04 (0.28)
  Left VLPFC Brain Activation | 0.02 (0.32) | 0.12 (0.44) | 0.07 (0.38) | 0.02 (0.23)
  Right DLPFC Brain Activation | 0.29 (0.32) | 0.32 (0.38) | 0.43 (0.37) | 0.39 (0.38)
  Right Caudate Brain Activation | 0.22 (0.34) | 0.16 (0.32) | 0.15 (0.52) | 0.19 (0.34)
  Right Putamen Brain Activation | 0.18 (0.28) | 0.16 (0.30) | 0.18 (0.36) | 0.15 (0.39)
  Right Dorsal ACC Activation | 0.03 (0.27) | 0.13 (0.32) | 0.09 (0.36) | 0 (0.25)
  Right VLPFC Brain Activation | 0.31 (0.25) | 0.34 (0.28) | 0.51 (0.30) | 0.40 (0.30)

5. Secondary Outcome: Stop Signal Reaction Time (SSRT)
Description: Behavioral performance on the stop signal task, as measured by stop signal reaction time calculated as mean go reaction time minus the stop-signal delay at 50% successful inhibition (SSD₅₀). Higher SSRT means longer latency before failed inhibition.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Standard Error); unit: Milliseconds
Groups:
- Participants With Bulimia Nervosa; Healthy Control Participants Without Bulimia Nervosa: Participants are scanned after 16 hours of fasting (Fasted Scan) on one day, and are scanned after a standardized meal on a separate day (Fed Scan). The order of these fasted and fed visits was counterbalanced across participants.
Arm/Group | Participants With Bulimia Nervosa | Healthy Control Participants Without Bulimia Nervosa
Number analyzed (Participants) | 28 | 28
Milliseconds
  Fasted Scan | 164.37 (16.31) | 151.70 (18.89)
  Fed Scan | 170.80 (79.14) | 166.58 (13.99)

6. Secondary Outcome: Stop Signal Task Inhibition
Description: Percent correct responses to stop trials on the Stop Signal Task measured by percent of stop trials on which participant successfully withheld a response (vs. failed to withhold response).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Standard Error); unit: percent correct responses
Arm/Group | Participants With Bulimia Nervosa | Healthy Control Participants Without Bulimia Nervosa
Number analyzed (Participants) | 28 | 28
percent correct responses
  Fasted Scan | 57.29 (2.00) | 55.56 (2.62)
  Fed Scan | 53.12 (3.05) | 56.25 (2.93)

ADVERSE EVENTS:
Time Frame: At baseline clinical interviews, the 16-hour fasting period before scan visits, and at the two scan visits (up to 3 weeks on average)
Arm/Group | Participants With Bulimia Nervosa | Healthy Control Participants Without Bulimia Nervosa
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 1/32 | 4/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Bulimia Nervosa (N=32) | Healthy Control Participants Without Bulimia Nervosa (N=32)
Reported Headache (Injury, poisoning and procedural complications) | 0 | 2 — Reported anticipated side effects from the fasting period
Potential structural abnormality identified on MRI (Nervous system disorders) | 1 | 2 — Incidental finding

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-05-01): https://cdn.clinicaltrials.gov/large-docs/57/NCT04409457/Prot_SAP_000.pdf
  • Informed Consent Form (2024-07-10): https://cdn.clinicaltrials.gov/large-docs/57/NCT04409457/ICF_001.pdf